CLINICAL TRIAL: NCT06052735
Title: Association Among Pain Perception, Severity of Temporomandibular Joint Dysfunction, and Spinal Health in Caregivers of Stroke Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Halime Arikan, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13.26
Record Dates: First submitted 2023-09-13; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Pain; Discomfort; Caregiver; Temporomandibular Disorder; Spine
Keywords: Caregiver; Pain; Discomfort; Spine; Temporomandibular disorder
MeSH Terms: conditions — Pain; Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Correlation arm (Other)
  Interventions: Other: Correlation research

INTERVENTIONS:
Other: Correlation research — The relationship among pain perception, temporomandibular disorder severity and spine health

SUMMARY:
This study aims to examine pain perception, temporomandibular disorder severity and spine health in caregivers of stroke patients.

DETAILED DESCRIPTION:
The sample of the study will consist of caregivers who reside in Tokat and Kırıkkale, are over 18 years old, care for an individual who has had a stroke and volunteer to participate in the study. Individuals will be contacted via social media, and squestionnaires will be administered face-to-face to those who agree to participate in the study. According to the G*Power analysis, if the sample size is α= 0.05, β= 0.80, acceptable correlation coefficient r= 0.70, and negligible correlation coefficient r= 0.20, 16 individuals are sufficient to measure the relationship between two parameters. Since the relationship between four parameters will be evaluated, a total of 64 individuals are required.

Data for the study will be collected face-to-face by individual researchers using data tools that individuals can fill in themselves. Data will be collected from individuals with The Centrality of Pain Scale, Discomfort Intolerance Scale, Spine Functional Index, and Fonseca Anamnestic Index instruments.

Statistical Package for Social Sciences (SPSS), version 22.0 computer package program for Windows, will be used for statistical analysis. Statistical data will be expressed as mean ± standard deviation (X±SD), median or percentage (%). One Sample Kolmogorov Smirnov test will be performed to show parametric or nonparametric distribution of the data. When parametric test assumptions are met, the relationship between parameters is determined by Spearman correlation test; When parametric test assumptions are not met, the relationship between the parameters will be examined with the Pearson correlation test. Statistical significance value will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* To be volunteer

Exclusion Criteria:

* Those who cannot speak, read or write Turkish.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
The Centrality of Pain Scale | up to 3 months
  The Centrality of Pain Scale will be used to assess pain perception. It is a 10-item questionnaire in which each item is rated on a 5-point Likert type (1: strongly disagree, 2: disagree, 3: neither agree nor disagree, 4: agree, 5: strongly agree). Items 2, 4, and 9 are reverse scored. The total score is the sum of all item scores. Higher scores reflect more "centralized" pain. The maximum score is 50, and the minimum score is 10. Turkish version, validity, and reliability study was conducted.
Discomfort Intolerance Scale | up to 3 months
  Tolerance to physical discomfort and pain will be evaluated with the Discomfort Intolerance Scale. The scale consists of 7-point Likert-type questions, and the answer options vary between 0 (not at all suitable for me) and 6 (completely suitable for me). Its Turkish version, validity, and reliability study is available.
Spine Functional Index | up to 3 months
  Spine Functional Index is a scale of 25 questions developed to examine the impact of spine-related symptoms on functionality. Each question is scored as 0, 0.5, and 1. The total score is calculated as a percentage, and a score approaching 100% indicates normal spinal functions. The Turkish version, validity, and reliability were tested.
Fonseca Anamnestic Index | up to 3 months
  The presence and severity of temporomandibular disorder in individuals will be evaluated with the Fonseca Anamnestic Index. The Fonseca Anamnestic Index consists of 10 questions. The participant is asked to answer each question as 'Yes' (10 points), 'No' (0 points), and 'Sometimes' (5 points). The questionnaire score is scored for all questions, and the severity of temporomandibular disorder is classified based on the total score: no temporomandibular disorder (0-15 points), mild temporomandibular disorder (20-40 points), moderate temporomandibular disorder (45-65 points), severe TMJD ( 70-100). The Turkish version, validity, and reliability were tested.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)